CLINICAL TRIAL: NCT02855203
Title: Stereotactic Radiotherapy and Anti-PD1 Antibody (Pembrolizumab) for Oligometastatic Renal Tumours
Acronym: RAPPORT
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Peter MacCallum Cancer Centre, Australia (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 15/143
Record Dates: First submitted 2016-07-28; First posted 2016-08-04 (Estimated); Results first posted 2023-08-03 (Actual); Last update posted 2023-08-03 (Actual); Status verified 2023-08

CONDITIONS: Renal Cell Carcinoma
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- SABR + Pembrolizumab (Experimental): SABR treatment (18Gy-20Gy/1#) followed by 200mg pembrolizumab IV once every 3 weeks for a total of 8 cycles
  Interventions: Radiation: Stereotactic Ablative Body Radiosurgery (SABR); Drug: Pembrolizumab

INTERVENTIONS:
Radiation: Stereotactic Ablative Body Radiosurgery (SABR) — 18-20Gy in 1 fraction
Drug: Pembrolizumab — Pembrolizumab at a dose of 200mg IV, 3-weekly will be delivered for a duration of 6 months, commencing 5 days (+/- 3 days) from the last dose of SABR.

SUMMARY:
This investigator driven study will examine the safety, efficacy and biological effects of combining pembrolizumab (MK-3475) an antibody targeted against anti-programmed cell death 1 (PD-1), with stereotactic ablative body radiotherapy (SABR) for oligometastatic renal cell carcinoma (RCC). The investigators hypothesise that the safety profile of this combination will be clinically acceptable.

DETAILED DESCRIPTION:
Dual institutional, single arm, unblinded, phase I/II study.

ELIGIBILITY:
Inclusion Criteria:

1. Has provided written informed consent for the trial.
2. Be at least 18 years of age on day of signing informed consent.
3. Have oligometastases (1-5 metastases), and measurable disease based on RECIST 1.1.
4. Participants must have a histologically or cytologically confirmed metastatic renal cell carcinoma. Oligometastatic lesions do not need to be biopsied but they must be clinically consistent to represent metastatic disease.
5. Patient can either be treatment naïve or have previously received up to 2 lines of systemic treatment (eg. Pazopanib or Sunitinib). The total number of metastases throughout the pre-trial period should not number more than 5.
6. Must have had surgical consideration for metastasectomy and thought appropriate for SABR due to medical inoperability, technical factors or patient declining surgery.
7. Must have at least one metastasis for which SABR is technically deliverable.
8. Be willing to provide archival tissue from a previously biopsied or excised primary or metastatic RCC lesion (if available). If safe to do so, a request for newly obtained specimen (obtained up to 4 weeks prior to initiation of treatment) will be made, however participation for this biopsy is entirely optional.
9. Have a performance status of 0-2 on the ECOG Performance Scale
10. Demonstrate adequate organ function as defined below all screening labs should be performed within 10 days of registration.

    * Absolute neutrophil count (ANC) - ≥1.5 X 10^9/L
    * Platelets - ≥100 X 10^9/L
    * Hemoglobin - ≥90 g/L or ≥5.6 mmol/L without transfusion or EPO dependency (within 7 days of assessment)
    * Serum creatinine OR Measured or calculated creatinine clearance (GFR can also be used in place of creatinine or CrCl) - ≤1.5 X upper limit of normal (ULN) OR ≥60 mL/min for participant with creatinine levels > 1.5 X institutional ULN
    * Serum total bilirubin - ≤ 1.5 X ULN OR Direct bilirubin ≤ ULN for participants with total bilirubin levels > 1.5 ULN
    * AST (SGOT) and ALT (SGPT) - ≤ 2.5 X ULN OR ≤ 5 X ULN for participants with liver metastases
    * Albumin - >2.5 mg/dL
    * International Normalized Ratio (INR) or Prothrombin Time (PT) - ≤1.5 X ULN unless participant is receiving anticoagulant therapy as long as PT or PTT is within therapeutic range of intended use of anticoagulants
    * Activated Partial Thromboplastin Time (aPTT) - ≤1.5 X ULN unless participant is receiving anticoagulant therapy as long as PT or PTT is within therapeutic range of intended use of anticoagulants
11. Life expectancy > 12 months.
12. Be willing and able to comply with all study requirements, including treatment, attending assessments and follow-up.
13. Female participant of childbearing potential should have a negative urine or serum pregnancy within 72 hours prior to receiving the first dose of study medication. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.
14. Female participants of childbearing potential should be willing to use 2 methods of birth control or be surgically sterile, or abstain from heterosexual activity for the course of the study through 120 days after the last dose of study medication (see Section 9.4.2: Contraception). Participants of childbearing potential are those who have not been surgically sterilized or have not been free from menses for > 1 year.
15. Male participants should agree to use an adequate method of contraception starting with the first dose of study therapy through 120 days after the last dose of study therapy

Exclusion Criteria:

1. Based on clinician assessment of disease volume and rate of progression of patient's tumor deposits, the patient requires immediate TKI therapy.
2. Has had previous high dose radiotherapy (biological equivalent of 30Gy in 10#) to an area to be treated which includes vertebral bodies (see below).

   Note: Previous high dose radiotherapy is defined as a biological equivalent dose to above that of 30 Gy in 10 fractions using an alpha/beta ratio [82] of 3. Where a patient has received radiotherapy to an equivalent or lower dose than defined above, stereotactic radiotherapy of the area may be considered. In doing so, assessment of the volume and total dose received by any overlap region must be made, and documented by generating a cumulative plan incorporating both the previous and current treatment fields. It is the treating radiation oncologist's responsibility to review both the current plan and the cumulative plan inclusive of previous radiotherapy.
3. Has evidence of untreated or active intracranial metastases. Patients who have had fully resected brain metastasis or those controlled by stereotactic radiotherapy are eligible as long as they are not requiring corticosteroids for symptomatic control.
4. Has evidence of Spinal Cord Compression.
5. Has a Spinal Instability Neoplastic Score ≥ 7 unless lesion reviewed by a neurosurgical service and considered stable (see Appendix 3).
6. Requires surgical fixation of bone lesion for stability. This must be performed before enrollment into the trial.
7. Has a diagnosis of immunodeficiency or is receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days of registration.
8. Has a known history of active TB (Bacillus Tuberculosis).
9. Hypersensitivity to pembrolizumab or any of its excipients.
10. Has had a prior anti-cancer monoclonal antibody (mAb) within 4 weeks of registration or who has not recovered (i.e., ≤ Grade 1 or at baseline) from adverse events due to agents administered more than 4 weeks earlier.
11. Has had prior chemotherapy, targeted small molecule therapy, or radiation therapy within 2 weeks of registration or who has not recovered (i.e., ≤ Grade 1 or at baseline) from adverse events due to a previously administered agent.

    Note: Participants with ≤ Grade 2 neuropathy are an exception to this criterion and may qualify for the study.

    Note: If participant received major surgery, they must have recovered adequately from the toxicity and/or complications from the intervention prior to starting therapy.
12. Has a known additional malignancy that is progressing or requires active treatment. Exceptions include basal cell carcinoma of the skin or squamous cell carcinoma of the skin that has undergone potentially curative therapy or in situ cervical cancer.
13. Has known active central nervous system (CNS) metastases and/or carcinomatous meningitis. Participants with previously treated brain metastases may participate provided they are stable (without evidence of progression by imaging for at least four weeks prior to the first dose of trial treatment and any neurologic symptoms have returned to baseline), have no evidence of new or enlarging brain metastases, and are not using steroids within 7 days of registration. This exception does not include carcinomatous meningitis which is excluded regardless of clinical stability.
14. Has active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (e.g. thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment.
15. Has known history of, or any evidence of active, non-infectious pneumonitis.
16. Has an active infection requiring systemic therapy.
17. Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the participant's participation for the full duration of the trial, or is not in the best interest of the participant to participate, in the opinion of the treating investigator.
18. Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
19. Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the screening visit through 120 days after the last dose of trial treatment.
20. Has received prior therapy with an anti-PD-1, anti-PD-L1, or anti-PD-L2 agent.
21. Has a known history of Human Immunodeficiency Virus (HIV) (HIV 1/2 antibodies).
22. Has known active Hepatitis B (e.g., HBsAg reactive) or Hepatitis C (e.g., HCV RNA [qualitative] is detected).
23. Has received a live vaccine within 30 days of registration

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2016-10-20 (Actual); Primary Completion 2020-05-22 (Actual); Study Completion 2020-05-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shankar Siva, Prof, Study Chair — Peter MacCallum Cancer Centre, Australia
Locations (2):
- Australia (2):
  - Princess Alexandra Hospital, Woolloongabba, Queensland
  - Peter MacCallum Cancer Centre, Melbourne, Victoria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Siva S, Bressel M, Wood ST, Shaw MG, Loi S, Sandhu SK, Tran B, A Azad A, Lewin JH, Cuff KE, Liu HY, Moon D, Goad J, Wong LM, LimJoon M, Mooi J, Chander S, Murphy DG, Lawrentschuk N, Pryor D. Stereotactic Radiotherapy and Short-course Pembrolizumab for Oligometastatic Renal Cell Carcinoma-The RAPPORT Trial. Eur Urol. 2022 Apr;81(4):364-372. doi: 10.1016/j.eururo.2021.12.006. Epub 2021 Dec 23. PMID 34953600
- [Derived] Pryor D, Bressel M, Lawrentschuk N, Tran B, Mooi J, Lewin J, Azad A, Colyer D, Neha N, Shaw M, Chander S, Neeson P, Moon D, Cuff K, Wood S, Murphy DG, Sandhu S, Loi S, Siva S. A phase I/II study of stereotactic radiotherapy and pembrolizumab for oligometastatic renal tumours (RAPPORT): Clinical trial protocol. Contemp Clin Trials Commun. 2021 Jan 6;21:100703. doi: 10.1016/j.conctc.2021.100703. eCollection 2021 Mar. PMID 33490707

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | SABR + Pembrolizumab
Started | 30
Completed | 30
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | SABR + Pembrolizumab
Number analyzed (Participants) | 30
Age, Continuous [Median (Full Range); unit: years] | 62 [47 to 80]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 23
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Toxicities Measured Using CTCAE Version 4.03
Description: Number of Participants with Grade 3 Treatment Related Adverse Events as determined using CTCAE version 4.03 criteria. This standard criteria can be found through National Cancer Institute (https://ctep.cancer.gov/protocoldevelopment/electronic_applications/ctc.htm). Grade 3 treatment-related events are high grade toxicities.
Time Frame: Up to 24 months after SABR treatment
Measure: Number; unit: participants with G3 TRAEs
Arm/Group | SABR + Pembrolizumab
Number analyzed (Participants) | 30
participants with G3 TRAEs | 4

2. Secondary Outcome: Overall Survival
Time Frame: From start of treatment until the date of death from any cause assessed up to 2 years
Measure: Number; unit: percentage of participants
Arm/Group | SABR + Pembrolizumab
Number analyzed (Participants) | 30
percentage of participants | 74

3. Secondary Outcome: Freedom From Local Progression (FFLP)
Description: Freedom from local progression (FFLP) was defined as the absence of progressive disease by the Response Evaluation Criteria in Solid Tumors criteria
Time Frame: From start of treatment until the date of first local progression or until the date of death from any cause, whichever occurs first, assessed up to 2 years
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | SABR + Pembrolizumab
Number analyzed (Participants) | 30
percentage of participants | 92 [80 to 97]

4. Secondary Outcome: Distant Progression Free Survival (DPFS)
Description: Percentage of Participants with Distant Progression Free Survival (DPFS)
Time Frame: From start of treatment until the date of first distant progression or until the date of death from any cause, whichever occurs first, assessed at 2 years
Measure: Number (95% Confidence Interval); unit: percentage of participants with DPFS
Arm/Group | SABR + Pembrolizumab
Number analyzed (Participants) | 30
percentage of participants with DPFS | 52 [33 to 69]

5. Secondary Outcome: Overall Response Assessed Using RECIST 1.1
Description: Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by CT: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR.
Time Frame: 24 months
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | SABR + Pembrolizumab
Number analyzed (Participants) | 30
percentage of participants | 63 [44 to 80]

6. Secondary Outcome: Pain Assessed Using the Numerical Pain Rating Scale
Description: The number of patients who reported a pain score >0 at least once after treatment. Numerical Pain Rating Score, 0-10 scale with 0 representing no pain, to 10 representing the worst possible pain.
Time Frame: From commencement of treatment up to 2 years.
Measure: Count of Participants; unit: Participants
Arm/Group | SABR + Pembrolizumab
Number analyzed (Participants) | 30
Participants | 22

ADVERSE EVENTS:
Time Frame: Up to 2 years
Arm/Group | SABR + Pembrolizumab
All-Cause Mortality (participants affected / at risk) | 7/30
Serious Adverse Events (participants affected / at risk) | 4/30
Other Adverse Events (participants affected / at risk) | 0/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | SABR + Pembrolizumab (N=30)
respiratory (Respiratory, thoracic and mediastinal disorders) | 4 — haemoptysis, pneumonitis, or dyspnoea, irrespective of relatedness or cause

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-01-16): https://cdn.clinicaltrials.gov/large-docs/03/NCT02855203/Prot_SAP_000.pdf